CLINICAL TRIAL: NCT05080634
Title: Analysis of Incidence and Risk Factors Associated With Gastroesophageal Reflux Disease and Esophagitis After Peroral Endoscopic Myotomy
Brief Title: Analysis of Prevalence and Risk Factors Associated With Gastroesophageal Reflux Disease and Esophagitis After Peroral Endoscopic Myotomy
Status: Recruiting | Type: Observational
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 22042020
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Achalasia; GERD
Keywords: Peroral endoscopic myotomy; High-resolution esophageal manometry
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients who underwent POEM — chalasia patients were recruited from a single center. The pre- and postoperative assessments included Eckardt scores, GerdQ questionnaire, high-resolution esophageal manometry, esophagogastroscopy and pH monitoring.

SUMMARY:
Achalasia is an uncommon disorder that results from the degeneration of ganglion cells of the myenteric plexus in the lower esophageal wall. Peroral endoscopic myotomy (POEM) is a minimally invasive procedure capable of overcoming limitations of achalasia treatments. This study aimed to: 1) identify the prevalence of reflux esophagitis and asymptomatic GERD in patients who underwent POEM, and 2) evaluate patient and intraprocedural variables associated with post-POEM GERD.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are 18 years of age and older and are willing to sign an Informed Consent Form (ICF)
2. Achalasia patients who underwent POEM

Exclusion Criteria:

1. Lack of written consent for participation in the study
2. Conditions which are contraindication to Esophagogastroscopy and High-resolution Esophageal Manometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated at a single center who had a complete GERD evaluation after POEM will be included in the study. Demographics, preoperative and follow-up data, results of functional studies and procedural data will be collected and analyzed.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of gastroesophageal reflux after peroral endoscopic myotomy (POEM) | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chaber-Ciopińska, PhD, Principal Investigator — The Maria Sklodowska-Curie National Research Institute of Oncology
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Poland